CLINICAL TRIAL: NCT03147209
Title: Pilot Intervention-Exercise for the Weight, Healthy Eating, and Exercise for the Long-Haul
Acronym: PIE WHEEL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never received funding.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Matthew Thiese, Assistant Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PPRT-2015-T1
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Obesity; Commercial Motor Vehicle Driver
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: This is a feasibility pilot study for a health coaching intervention for truck drivers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Coaching (Experimental): This group will undergo coaching and activities to improve strength and balance.
  Interventions: Behavioral: Health Coaching

INTERVENTIONS:
Behavioral: Health Coaching — This intervention will consist of health coaching, goal setting and self directed activities to improve strength and balance.

SUMMARY:
Truckers face many unique challenges in their work that may adversely impact their health, including time constraints, sedentary job tasks, and a 'moving-workplace' environment with associated limitations to access healthy food and safe places to be physically active. These issues make it difficult to form and maintain healthy lifestyle habits and contribute to the high prevalence of injuries from both crashes and falls among truckers is supported by an increase in obesity among truckers with longer durations of employment.

The investigators propose to develop and pilot test the Exercise Intervention of the Worksite Health, Eating and Exercising for the Long-haul (WHEEL)'s weight loss intervention. This pilot exercise intervention is aimed at achieving meaningful improvement in grip strength, balance, and gait over 6 weeks. The investigators will use pilot sample of 15 obese (BMI ≥ 30 kg/m2) truckers, documenting changes in these measures. Individualized assessments will be utilized. The investigators will aim to complete the following:

1. Evaluate the feasibility of the PIE WHEEL intervention for CMV drivers will result in greater strength comparing baseline with 6 week outcomes.

   1. Determine the extent to which drivers will participate in PIE WHEEL
   2. Determine the extent of change in strength, balance and gait realized by PIE WHEEL participation
2. Evaluate safety events (crashes, near misses, falls) in the week prior to PIE WHEEL and the final week of PIE WHEEL a. Solicit driver perceptions of their own safety of ingress and egress related to PIE WHEEL participation

DETAILED DESCRIPTION:
Commercial Motor Vehicle Drivers (CMV Drivers), also known as truck drivers, face many unique challenges in their work environment that adversely impact their health, particularly obesity. Obesity is significantly related to CMV driver occupational injuries and deaths from crashes.1, 2 CMV Driver's challenges include time constraints, limited space inside the truck, mostly sedentary job tasks, poor access for parking large trucks, and a 'moving-workplace' environment. This environment has poor access to inexpensive, ready-to-eat, healthy food and places for exercising and showering. These constraints make it difficult to form and maintain healthy lifestyle habits. That these influences likely contribute to the disproportionately high prevalence of obesity among CMV drivers is supported by an increase in obesity among truckers with longer durations of employment.3

Prior efforts to reduce obesity were not successful for trucking.4-7 However two, short-term pilot studies showed promise utilizing motivational interviewing in achieving a 3.5 kg weight loss.8, 9 Accordingly, development of interventions is needed to improve CMV driver's health and safety through weight loss by helping the truck driver's change his/her response to the unique challenges of their work environment.

Herein, The investigators propose the pilot intervention-exercise (PIE) aspect of the Worksite Health, Eating and Exercising for the Long-haul (WHEEL), a behavior-based intervention. The PIE WHEEL will assess the feasibility, acceptability and potential safety improvements of an exercise intervention on quantifiable outcomes that impact workers compensation concerns including musculoskeletal disorders and slips, trips and falls.

PIE WHEEL will utilize health coaches to deliver an intervention using individual goal setting to establish behaviors (exercise only for this pilot study) known to be associated with successful weight loss and/or weight loss maintenance and subsequent safety outcomes designed to meet the challenges of CMV drivers. The investigators will enroll 15 participants for a 6 week exercise intervention.

SPECIFIC AIMS

1. Evaluate the feasibility of the PIE WHEEL intervention for CMV drivers will result in greater strength comparing baseline with 6 week outcomes.

   1. Determine the extent to which drivers will participate in PIE WHEEL
   2. Determine the extent of change in strength, balance and gait realized by PIE WHEEL participation
2. Evaluate safety events (crashes, near misses, falls) in the week prior to PIE WHEEL and the final week of PIE WHEEL a. Solicit driver perceptions of their own safety of ingress and egress related to PIE WHEEL participation

Safety events (crashes and falls) are a meaningful outcomes in the transportation industry. Some of the causal factors related to these, including strength, vigilance, cardiovascular disease and obesity, may be influences by the PIE WHEEL intervention. This is compounded by the high obesity prevalence, which exceeds >65%, among truckers.10, 11 The personal and public health threat of obesity-related problems among truckers that includes falls and severe injuries are substantial and require intensive intervention efforts to reduce obesity. The investigators propose the PIE WHEEL intervention; a behavior based individualized exercise intervention utilizing health coaches to direct individual goal setting to address this need. This proposal is in direct response to comments from an unfunded R01 intervention that proposed both diet and exercise intervention for weight reduction. The assessment of feasibility, acceptance, and quantification of changes will further strengthen the R01 at the time of resubmission.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI>30kg/m2)
* Working as a commercial motor vehicle driver

Exclusion Criteria:

* unable to perform intervention (health coaching and goal setting

Ages: 21 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Improved Strength | 6 weeks
  Strength testing will be performed and changes in strength will be evaluated at baseline and after 6 weeks
Improved Balance | 6 weeks
  Balance testing will be performed and changes in balance will be evaluated at baseline and after 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No